CLINICAL TRIAL: NCT02625441
Title: A Randomized Phase III Study Comparing Trastuzumab, Pertuzumab Plus Docetaxel (TPD) Followed by 3 Cycles of Chemotherapy to the Current Standard Regimen as the Treatments of Early Breast Cancer
Brief Title: Adjuvant Trastuzumab, Pertuzumab Plus Docetaxel in the Treatment of Early HER2-positive Breast Cancer
Acronym: BOLD-1
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Heikki Joensuu, Professor, Research Director, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FBCG-01-2015; 2015-002323-25 (EudraCT Number)
Record Dates: First submitted 2015-12-05; First posted 2015-12-09 (Estimated); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer
Keywords: Breast cancer; docetaxel; pertuzumab; trastuzumab; HER2
MeSH Terms: conditions — Breast Neoplasms | interventions — pertuzumab; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Short anti-HER2 treatment (Experimental): Pertuzumab 840 mg, i.v., then 420 mg i.v., 3-weekly for 3 cycles; Trastuzumab 8 mg/kg, i.v., then 6 mg/kg, 3-weekly for 3 cycles; Docetaxel 75 mg/m2, i.v., 3-weekly for 3 cycles
  Interventions: Drug: Pertuzumab
- Standard anti-HER2 treatment (Active Comparator): Trastuzumab 8 mg/kg, i.v., then 6 mg/kg, 3-weekly for 3 cycles; Docetaxel 75 mg/m2, i.v., 3-weekly for 3 cycles; Trastuzumab 6 mg/kg, i.v., 3-weekly for for a total duration of one year
  Interventions: Drug: Trastuzumab

INTERVENTIONS:
Drug: Pertuzumab — Pertuzumab 420 mg i.v. 3-weekly for 3 cycles
  Other Names: Perjeta
  Arms: Short anti-HER2 treatment
Drug: Trastuzumab — Trastuzumab 6 mg/kg, i.v., 3-weekly for for a total duration of one year
  Other Names: Herceptin
  Arms: Standard anti-HER2 treatment

SUMMARY:
This randomized clinical trial compares two systemic treatments for HER2-positive breast cancer. The treatments are given either prior to breast surgery (as neoadjuvant treatment) or after breast surgery (as adjuvant treatment). In the investigational group (Group A) the study participants will receive a combination of two drugs directed at HER2 (two anti-HER2 antibodies) plus a chemotherapy agent (docetaxel) for a brief duration, and the patients allocated to the comparator group (Group B) will be treated with chemotherapy plus one anti-HER2 treatment (trastuzumab) for one year.

DETAILED DESCRIPTION:
In this study, patients who have been diagnosed with HER2-positive early breast cancer will be randomly allocated in a 1:1 ratio to receive either three 3-weekly cycles of trastuzumab, pertuzumab and docetaxel (TPD) for a total duration of 9 weeks, followed by three further cycles of chemotherapy (Group A) or three 3-weekly cycles of trastuzumab and docetaxel (TD) followed by three further cycles of chemotherapy and single-agent anti-HER2 antibody treatment to complete one year of anti-HER2 treatment (Group B). These systemic treatments may be administered either prior to breast surgery (as neoadjuvant treatment) or after breast surgery (as adjuvant treatment). The study participants are required to have histologically verified breast cancer with a moderate to high risk for breast cancer recurrence despite macroscopically complete surgery for the breast tumor. The moderate/high risk of breast cancer recurrence is defined by presence of cancer in the axillary lymph nodes, or if the axillary lymph nodes do not contain cancer, by presence of a tumor larger than one centimeter in the breast. The study patients are followed up during the study treatments and after their completion with physical examination, blood tests, cardiac tests and, whenever indicated, with imaging. Approximately 520 patients will be randomly allocated to each of the two groups. The study hypothesis is that the regimen containing TPD may be more effective than the Group B treatment despite its brief duration.

ELIGIBILITY:
Inclusion Criteria:

* Patient has provided a written informed consent prior to study-specific screening procedures, with the understanding that she has the right to withdraw from the study at any time, without prejudice.
* Woman > 18 years of age.
* Histologically confirmed invasive breast cancer.
* HER2-positive breast cancer (preferably assessed with in situ hybridization; CISH, FISH or SISH; if not available with immunohistochemistry 3+)
* A high risk of breast cancer recurrence with one of the following: i) Pathological N0 with the longest invasive tumor diameter >10 mm; ii) Histologically confirmed regional node positive disease

Exclusion Criteria:

* Presence of distant metastases.
* Inflammatory breast cancer.
* Clinically significant (i.e. active) cardiac disease (e.g. congestive heart failure, symptomatic coronary artery disease and cardiac arrhythmia not well controlled with medication) or myocardial infarction within the last 12 months.
* Left ventricular ejection fraction less than 50% (or under the institutional normal reference range) assessed by echocardiography or isotope cardiography.
* ER and HER-2 status (via in situ hybridization or immunohistochemistry) not determined.
* The WHO performance status > 1.
* Pregnant or lactating women.
* Women of childbearing potential unless using a reliable and appropriate contraceptive method. Women must have been amenorrheic for at least 12 months prior to study entry to be considered postmenopausal and to have no childbearing potential. Women of childbearing potential (menstruating within 12 months of study entry), or with no hysterectomy and age < 55, must have a negative pregnancy test at baseline.
* Randomization more than 12 weeks after the date of breast surgery.
* Organ allografts with immunosuppressive therapy required.
* Major surgery (except breast surgery) within 4 weeks prior to study treatment start, or lack of complete recovery from the effects of major surgery.
* Participation in any investigational drug study within 4 weeks preceding treatment start.
* Patients with a history of uncontrolled seizures, central nervous system disorders or psychiatric disability judged by the investigator to be clinically significant precluding study participation.
* Multifocal breast cancer when the largest cancer focus is not HER2-positive.
* History of another malignancy or contralateral invasive breast cancer within the last five years except cured basal cell carcinoma of skin or carcinoma in situ of the uterine cervix (exception: patients with bilateral HER2-positive breast cancer are eligible).
* One or more of the following: Blood hemoglobin < 10.0 g/dL, neutrophils < 1.5 x 109/L; platelet count < 120 x 109/L; Serum/plasma creatinine > 1.5 x Upper Limit of Normal (ULN); Serum/plasma bilirubin > ULN; Serum/plasma ALT and/or AST > 1.5 x ULN; Serum/plasma alkaline phosphatase > 2.5 x ULN
* Serious uncontrolled infection or other serious uncontrolled concomitant disease.
* Unwilling or unable to comply with the protocol for the duration of the study.
* History of hypersensitivity to the investigational products or to drugs with similar chemical structures.
* Pre-existing motor or sensory neurotoxicity of a severity ≥ grade 2 by CTCAE version 4, unless related to mechanical etiology.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 516 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Invasive disease-free survival | 7 years
  Time from the date of randomization to cancer recurrence or death.

SECONDARY OUTCOMES:
Overall survival | 7 years
  Time from the date of randomization to death.
Distant disease-free survival | 7 years
  Time from the date of randomization to distant recurrence of cancer or to death.
Left ventricle ejection fractions | 3 years
  Cardiac ejection fraction measured with echocardiography or isotope cardiography.
Adverse events of the treatments | 7 years
  Adverse events considered to be related to the treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Heikki Joensuu, M.D., Principal Investigator — Helsinki University Central Hospital
Locations (1):
- Helsinki University Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No